CLINICAL TRIAL: NCT03712839
Title: Cognitive and Cerebral Mechanisms of Anosognosia in Patients With Acquired Brain Damage: New Evaluation Strategies Based on Daily Tasks
Brief Title: Cognitive-functional Evaluation of Anosognosia
Status: Completed | Type: Observational
Sponsor: María Rodríguez Bailón (Other)
Collaborators: Universidad de Granada (Other)
Responsible Party: Sponsor-Investigator, María Rodríguez Bailón, Professor, University of Malaga
Organization: University of Malaga (Other)
Other Study IDs: PSI2016-80331-P
Record Dates: First submitted 2018-09-08; First posted 2018-10-19 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Anosognosia; Brain Damage
Keywords: Activities of Daily Living (ADL); Executive Deficit; Monitoring; Self Awareness
MeSH Terms: conditions — Agnosia; Brain Injuries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Acquired Brain Injury group with anosognosia: People with presence of an acquired brain damage and cognitive deficits relative to executive functions and memory. To determine the presence of anosognosia, patients must present an overestimation value of their capacities greater than 5 (>5) in the discrepancy index on the Patient Competency Rating Scale (PCRS) (Prigatano et al., 1998).
  Interventions: Other: Cognitive-functional evaluation
- Acquired Brain Injury group without anosognosia: People with presence of an acquired brain damage and cognitive deficits relative to executive functions and memory. These patients must present a score of < 5 on the PCRS Scale.
  Interventions: Other: Cognitive-functional evaluation
- Control group: Healthy participants matched in age, gender and educational level with the others two groups.
  Interventions: Other: Cognitive-functional evaluation

INTERVENTIONS:
Other: Cognitive-functional evaluation — The participants will be evaluated with a set of tools within the context of meaningful ADL.

SUMMARY:
Acquired brain damage patients usually show severe cognitive deficit that alter their performance on every day life activities. Some of them suffer anosognosia and they are not aware of their own limitations. This situation increases disability by producing a large number of unsafe behaviours, caregivers burn-out and impede rehabilitation by affecting patients desire to follow treatment instructions. From disciplines like Neuropsychology, Cognitive Neuroscience or Occupational Therapy, it is considered a crucial issue to investigate the cognitive and neural mechanisms responsible of anosognosia, as well as to increase our knowledge about the most efficient treatments to deal with this phenomenon. The main general objective of this project is to generate and validate a detailed cognitive assessment protocol within the context of ADL to evaluate the different cognitive components of consciousness proposed on the Toglia and Kirk´s model: 1) Offline componente: metacognitive knowledge and 2) Online component: emergent awareness, self-regulation, anticipatory awareness, self-evaluation and updating processes).

DETAILED DESCRIPTION:
The proposed protocol is composed by two ecological tools: The Cog-Awareness ADL Scale (ADL scale of metacognitive knowledge) and the Basic and Instrumental ADL performance based test (Awareness ADL), to identify the presence of cognitive deficits and anosognosia in patients with ABI always within the context of everyday life activities. One first specific aim is to test the convergent validity of the two proposed ecological tools with other traditional and validated measures usually used to assess similar cognitive processes and components of self-awareness. The second specific objective is to investigate the external validity of the ecological tools, by testing whether they are able to discriminate between acquired brain damage patients with and without anosognosia and a group of neurologically healthy participants on every component.

After conducting a literature review of the subject we found that this would be the first protocol developed to identify all these components in the same study.

ELIGIBILITY:
Inclusion Criteria:

* Presence of an acquired brain damage objectively observed with medical reports.
* Cognitive deficits relative to executive functions and/or memory evaluated by the team of professionals who recruit participants in the hospital.

Exclusion Criteria:

* Presence of a serious visuoperceptual deficit that makes it difficult to complete the ADL tasks, evaluated by the team of professionals who recruit participants in the hospital.
* Presence of an understanding deficit (aphasia) evaluated by the team of professionals who recruit participants in the hospital.
* Presence of spatial neglect evaluated with line cancellation and line bisection tests.
* Presence of motor deficits in both upper limbs that impedes to complete the ADL tasks.
* Total score in MMSE<18

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Acquired brain damage patients will be recruited on the collaborating hospitals and on different acquired brain damage organisations. Both, patients and control subjects, will be recruited from Málaga and Granada.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2016-10-18 (Actual); Primary Completion 2020-03 (Actual); Study Completion 2022-06 (Actual)

PRIMARY OUTCOMES:
The awareness ADL | 30-45 minutes
  Participants will be asked to do activities of daily living such as preparing a breakfast or dressing in which measures that evaluate components of anosognosia will be used. In the tasks of ADL conflict situations (and standardized solutions previously defined) and distractor objects will be presented. The total errors committed will be analyzed, as well as those committed only by conflict situations and distractor objects. The percentage of errors detected and corrected errors will be calculated.
  In addition, anticipatory awareness, self-evaluation and updating processes will be examined.
The Cog-Awareness ADL Scale | 10-15 minutes
  For the aim of this study, the Cog-Awareness ADL Scale, will have two versions, one to be administered to a direct caregiver and the other to the patient to observe the discrepancy index in relation to functionality-cognition. This tool allow to evaluate eight key cognitive abilities-task: manipulation difficulties, action schema, distraction, substitution, repetition, error detection, problem solving and task self-initiation in the two basic ADL and in the two instrumental ADL (BADL and IADL, respectively) (34 items). Both patients and caregivers must answer how often the patients present this cognitive-functional error in each of the 4 ADLs: 1: never, 2: sometimes, 3: quite often and 4: always. Two indices are calculated, one for BADL and one for IADL, adding all the scores of the two activities of each category among the number of activities answered. Lower punctuation is interpreted with worse results. There are 3 items that your scores should be reversed.

SECONDARY OUTCOMES:
Mini-Mental State Examination | 10 minutes
  General cognitive status. MMSE is a 30-point questionnaire that is used extensively in clinical and research settings to measure cognitive impairment. It is commonly used in medicine and allied health to screen for dementia. It is also used to estimate the severity and progression of cognitive impairment and to follow the course of cognitive changes in an individual over time; thus making it an effective way to document an individual's response to treatment.
Line cancellation test | 3-5 minutes
  General cognitive status. In the LCT the patient is asked to cross out all the lines (or particular items) on a sheet.
Line bisection test | 3-5 minutes
  General cognitive status. The LBT is a quick measure to detect the presence of unilateral spatial neglect (USN). To complete the test, one must place a mark with a pencil through the center of a series of horizontal lines. Usually, a displacement of the bisection mark towards the side of the brain lesion is interpreted as a symptom of neglect.
Key search test | 2-4 minutes
  Executive functions. Participants are required to search for an imaginary key they have lost on a field (a square on a piece of paper). By drawing their search route, an indication of search strategy and planning ability can be deduced.
INECO Frontal Screening | 6-10 minutes
  Executive functions. This screening test was designed to provide health professionals with a sensitive and specific executive screening test to determine frontal dysfunction in patients with dementia.
Color trail making | 6 minutes
  Executive functions. Numbered circles are printed with vivid pink or yellow backgrounds that are perceptible to colorblind individuals. For Part 1, the respondent uses a pencil to rapidly connect circles numbered 1-25 in sequence. For Part 2, the respondent rapidly connects numbered circles in sequence, but alternates between pink and yellow. The length of time to complete each trial is recorded, along with qualitative features of performance indicative of brain dysfunction, such as near-misses, prompts, number sequence errors, and color sequence errors.
Rey Auditory Verbal Learning Test | 10-15 minutes
  Semantic and episodic memory. The RAVLT evaluates a wide diversity of functions: short-term auditory-verbal memory, rate of learning, learning strategies, retroactive, and proactive interference, presence of confabulation of confusion in memory processes, retention of information, and differences between learning and retrieval.
Patient Competency Rating Scale | 6-10 minutes
  Metacognitive knowledge. The primary purpose of the PCRS is to evaluate self-awareness (the ability to appraise one's current strengths and weaknesses) following traumatic brain injury. The PCRS is a 30-item self-report instrument which asks the subject to use a 5-point Likert scale to rate his or her degree of difficulty in a variety of tasks and functions. The subject's responses are compared to those of a significant other (a relative or therapist) who rates the subject on the identical items. Impaired self-awareness may be inferred from discrepancies between the two ratings, such that the subject overestimates his/ her abilities compared to the other informant. Awareness of deficit may also be examined separately for activities of daily living, behavioral and emotional function, cognitive abilities, and physical function. Range Discrepancy index range 1-150.
  Mean healthy subjects: 144 range (120-150) and relatives 145 (range 134-150) (Prigatano, 1998)
Verbal Fluency Test | 5 minutes
  In this test the participants have to produce as many words as possible from a category in a 60 seconds. This category is semantic (animals) and phonemic, including words beginning with F, A and S.
Weekly Calendar Planning Activity (WCPA) | 20 minutes
  This is a performance based test that measures different executive functions, among which are: planning, problem solving, inhibition of non-relevant information and maintenance and monitoring of rules. In its short version, it is based on asking the patient to schedule 10 appointments (that appear in random order) during a 1 week span. Some appointments are incompatible with others, so the patient has to take them into account to plan correctly. In addition, the patient is asked to comply with 5 rules which are informed at the beginning of the test and are kept in view throughout the task. The test provides different variables for its analysis, as well as the successes when planning, such as the types of mistakes made, the ability to detect them, the time, the rules followed or the strategies used.

CONTACTS AND LOCATIONS:
Overall Officials: María Jesús Funes-Molina, Professor, Principal Investigator — Facultad de Psicología (Departamento de Psicología Experimental) - Campus de Cartuja s/n, Granada, 18071

REFERENCES:
- [Background] Folstein MF, Folstein SE, McHugh PR. "Mini-mental state". A practical method for grading the cognitive state of patients for the clinician. J Psychiatr Res. 1975 Nov;12(3):189-98. doi: 10.1016/0022-3956(75)90026-6. No abstract available. PMID 1202204
- [Background] Giovannetti T, Libon DJ, Hart T. Awareness of naturalistic action errors in dementia. J Int Neuropsychol Soc. 2002 Jul;8(5):633-44. doi: 10.1017/s135561770280131x. PMID 12164673
- [Background] Prigatano GP, Bruna O, Mataro M, Munoz JM, Fernandez S, Junque C. Initial disturbances of consciousness and resultant impaired awareness in Spanish patients with traumatic brain injury. J Head Trauma Rehabil. 1998 Oct;13(5):29-38. doi: 10.1097/00001199-199810000-00005. PMID 9753533
- [Background] Forde EM, Humphreys GW, Remoundou M. Disordered knowledge of action order in action disorganisation syndrome. Neurocase. 2004 Feb;10(1):19-28. doi: 10.1080/13554790490960459. PMID 15849156
- [Background] Schmidt J, Fleming J, Ownsworth T, Lannin NA. Video feedback on functional task performance improves self-awareness after traumatic brain injury: a randomized controlled trial. Neurorehabil Neural Repair. 2013 May;27(4):316-24. doi: 10.1177/1545968312469838. Epub 2012 Dec 27. PMID 23270921
- [Background] Rodriguez-Bailon M, Montoro-Membila N, Garcia-Moran T, Arnedo-Montoro ML, Funes Molina MJ. Preliminary cognitive scale of basic and instrumental activities of daily living for dementia and mild cognitive impairment. J Clin Exp Neuropsychol. 2015;37(4):339-53. doi: 10.1080/13803395.2015.1013022. Epub 2015 Mar 25. PMID 25805061
- [Background] Forde EM, Humphreys GW. Dissociations in routine behaviour across patients and everyday tasks. Neurocase. 2002;8(1-2):151-67. doi: 10.1093/neucas/8.1.151. PMID 11997493
- [Background] Sirigu A, Zalla T, Pillon B, Grafman J, Agid Y, Dubois B. Selective impairments in managerial knowledge following pre-frontal cortex damage. Cortex. 1995 Jun;31(2):301-16. doi: 10.1016/s0010-9452(13)80364-4. PMID 7555008
- [Background] Sirigu A, Zalla T, Pillon B, Grafman J, Agid Y, Dubois B. Encoding of sequence and boundaries of scripts following prefrontal lesions. Cortex. 1996 Jun;32(2):297-310. doi: 10.1016/s0010-9452(96)80052-9. PMID 8800616
- [Background] Torralva T, Roca M, Gleichgerrcht E, Lopez P, Manes F. INECO Frontal Screening (IFS): a brief, sensitive, and specific tool to assess executive functions in dementia. J Int Neuropsychol Soc. 2009 Sep;15(5):777-86. doi: 10.1017/S1355617709990415. Epub 2009 Jul 28. PMID 19635178
- [Background] Toglia J, Kirk U. Understanding awareness deficits following brain injury. NeuroRehabilitation. 2000;15(1):57-70. PMID 11455082
- [Derived] Merchan-Baeza JA, Rodriguez-Bailon M, Ricchetti G, Navarro-Egido A, Funes MJ. Awareness of cognitive abilities in the execution of activities of daily living after acquired brain injury: an evaluation protocol. BMJ Open. 2020 Oct 26;10(10):e037542. doi: 10.1136/bmjopen-2020-037542. PMID 33109646